CLINICAL TRIAL: NCT00566592
Title: The Effect of Ethanol on Overnight Glucose Regulation in Type 2 Diabetes Mellitus
Brief Title: The Effect of Ethanol on Overnight Glucose Regulation in Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mark Burge, Professor of Medicine, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: DK61990 (completed); DK061990
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes, Insulin Requiring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ethanol; Carbonated Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Oral ethanol, overnight
  Interventions: Other: oral ethanol, overnight
- 2 (Experimental): IV ethanol, overnight
  Interventions: Other: IV ethanol
- 3 (Placebo Comparator): Placebo, overnight
  Interventions: Other: soda water
- 4 (Placebo Comparator): Placebo, daytime
  Interventions: Other: soda water

INTERVENTIONS:
Other: oral ethanol, overnight — Oral ethanol before bedtime to achieve approximate BAL of 0.08%
  Arms: 1
Other: IV ethanol — IV ethanol before bedtime to achieve approximate BAL of 0.08%
  Arms: 2
Other: soda water — Oral Placebo before bedtime to achieve approximate BAL of 0.00%
  Arms: 3
Other: soda water — Oral Placebo to achieve approximate daytime BAL of 0.00%
  Arms: 4

SUMMARY:
Hypoglycemia is the principal barrier to the achievement of target glycemic goals in type 2 diabetes. Alcohol consumption is very prevalent in our society and a proven cause of hypoglycemia. Population studies suggest that elderly, insulin requiring type 2 diabetes patients are particularly vulnerable to severe hypoglycemia and that this problem accounts for an estimated $50 million or more in healthcare costs in the USA each year. We hypothesize that low dose ethanol significantly increases the vulnerability to overnight hypoglycemia and impairs the recovery of plasma glucose in elderly, insulin requiring patients with type 2 diabetes. Our preliminary studies suggest that low dose ethanol impairs recovery from day time insulin-induced hypoglycemia in type 2 diabetes patients but not in age matched healthy control subjects. The proposed studies will examine the effects of low dose ethanol on overnight glucose regulation in elderly, insulin requiring type 2 diabetes patients and will establish the mechanism of these impairments through a series of systematic evaluations. Specifically, these studies will document suppression of the dawn phenomenon by ethanol, and/or exacerbation of a deficient counterregulatory response to hypoglycemia during sleep, especially growth hormone. Specific mechanisms for the suppression of growth hormone to be examined include that evening ethanol (3) inhibits peak overnight ghrelin secretion and/or (4) reduces pituitary sensitivity to GHRH. Additionally, these studies will characterize (5) the dose response characteristics of ethanol on overnight glucose homeostasis and will (6) carefully evaluate the effect of the timing of ethanol administration in relation to meal ingestion on overnight hypoglycemic vulnerability. To address these aims, we will assess the effect of moderate doses of orally administered ethanol or placebo on overnight growth hormone release, ghrelin, total IGF-1, free IGF-1, insulin-like growth factor binding protein 1 (IGFBP-1) concentrations, glucose production and other parameters of glucose homeostasis among elderly control subjects versus elderly, insulin requiring subjects with type 2 diabetes. These important studies will provide a scientific basis for the prevention of overnight hypoglycemia (and the attendant cost savings) by providing mechanistic insights into the causes of nocturnal hypoglycemia.

ELIGIBILITY:
Inclusion Criteria: All type 2 diabetes subjects will be aged 50 to 75 years and will have carried the diagnosis of diabetes according to standard criteria and will be receiving insulin therapy alone or in combination with oral diabetes medications for at least 6 months. To exclude subjects with type 1 diabetes, all patients will be anti-GAD antibody negative and will retain the ability to secrete some nominal level of c-peptide in response to stimulation (i.e.- at least 2 ng/ml after ingesting Boost Plus). All subjects will be mentally fit to give informed consent. Nondiabetic control subjects will meet similar inclusion criteria (except for diabetes and hemoglobin A1C criteria). Control subjects will be matched as a group for age, gender and BMI. Finally, control subjects will undergo a standard 75 gram Oral Glucose Tolerance Test to assure the presence of normal glucose tolerance (142).

Exclusion Criteria: Exclusion criteria for all study subjects will include the existence of severe cardiovascular, hepatic or renal disease, or current malignancy as determined by the screening evaluation. Subjects with a past or current history of drug or alcohol abuse will also be excluded from study, as will subjects with a previously diagnosed seizure disorder, subjects with sleep apnea by medical history or as demonstrated during the accommodation sleep study night, subjects with diabetic gastroparesis, or subjects receiving current treatment medications that interfere with glucose homeostasis other than for diabetes therapy (e.g.- glucocorticoids, orlistat). Because of the known adverse effects of ethanol on unborn children, current intrauterine pregnancy will exclude patients from study. A body mass index greater than 36 kg/m2 will also be exclusionary. Additionally, subjects with a score of more than eight points on the Alcohol Use Disorders Identification Test (AUDIT) will be excluded from study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Rate of glucose recovery from hypoglycemia. | Hours

SECONDARY OUTCOMES:
Hormone and substrate concentrations | Hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Burge, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Clincal and Translational Science Center, Albuquerque, New Mexico, United States